CLINICAL TRIAL: NCT05669053
Title: Evaluating the Effectiveness of a Roblox Video Game for Children and Adolescents to Improve Body Image: Randomised Controlled Trial
Brief Title: The Impact of Playing Super U on Pre-adolescents' Body Image
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Collaborators: Unilever R&D (Industry); C+R research agency (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HAS.22.11.040
Record Dates: First submitted 2022-12-14; First posted 2022-12-30 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Body Image

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The datasets given to the statistician will be blinded to the condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Super U Story intervention (Experimental): Participants in this condition will be asked to play the Roblox video game, Super U Story with the goal of reaching the end of the game (approximately 20-30 minutes)
  Interventions: Behavioral: Super U Story intervention
- Alternative Roblox game (Active Comparator): Participants in this condition will be asked to play the Roblox video game, Rainbow Friends Story (Color Story) with the goal of reaching the end of the game (approximately 20-30 minutes)
  Interventions: Behavioral: Alternative Roblox game
- Online word search (Active Comparator): Participants in this attention control condition will be asked to complete as many online word searches on the topic of animals as they can in 20-30 minutes.
  Interventions: Behavioral: Online word search

INTERVENTIONS:
Behavioral: Super U Story intervention — Participants in this condition will be asked to play a Roblox adventure video game called 'Super U Story'. They will play the game once and have between 6 - 30 minutes to complete the game.
  Arms: Super U Story intervention
Behavioral: Alternative Roblox game — Participants in this condition will be asked to play an alternative Roblox adventure video game called Rainbow Friends Story (colour story). They will play the game once and have between 6 - 30 minutes to complete the game.
  Arms: Alternative Roblox game
Behavioral: Online word search — Participants in this condition will have 20 minutes to complete a series of word searches online.
  Arms: Online word search

SUMMARY:
Body image concerns can have serious physical and psychological consequences on young people, including anxiety, depression, risk taking behaviours, eating disorders and suicidal ideation.

Micro-interventions (brief, low intensity interventions), offer an alternative to traditional, intense interventions that aim to immediately improve specific symptoms. Body image micro-interventions have proven effective at providing immediate and short-term improvements in body image among adolescents within digital and community settings. To date, utilising micro interventions in the world of gaming remains unexplored. Specifically, the Roblox platform which is hugely popular among young people (Roblox, September 2022).

As such, the aim of the present study is to conduct a randomised controlled trial (RCT) to evaluate the immediate and short-term impact of a Roblox game, Super U story, on American children and adolescents' body image, mood, internalisation of appearance ideals and social media literacy. The primary outcome is immediate change in state-based body satisfaction. Secondary outcomes include immediate changes in state-based mood and body functionality and short-term changes in trait body esteem, body appreciation, internalisation of appearance ideals and social media literacy.

The Super U story was developed through a collaboration between Dove (Unilever), Toya (game developers) and The Centre for Appearance Research. It was specifically designed to target sociocultural risk and protective factors for body image including social media literacy, appearance comparisons, positive body image and teasing/bullying around appearance.

The comparison control conditions include an active control; an alternative Roblox game; Rainbow Friends story which has been matched to the intervention on style, length, and age appropriateness (omitting body image messaging) and an attention control whereby participants complete a series of word searches.

To undertake the main trial, 1,479 girls and boys will be recruited through an external research agency. Participants will be randomised to one of three conditions: 1) the Super U story intervention, 2) alternative Roblox game or 3) attention control. All participants will be encouraged to play the game/word search for a maximum of 30 minutes, where they will be assessed on state-body image and mood immediately before and after completing the game/word search. All participants will be assessed on trait body esteem, body appreciation, internalisation of appearance ideals and social media literacy at baseline (one week pre-intervention) and again at one-week post intervention.

At the end of the study, all participants will receive a debrief form, outlining the study aims and objectives, and additional resources for body and eating concerns.

DETAILED DESCRIPTION:
Background:

Extensive research has established that body image issues are evident in early adolescence and can have far-reaching negative consequences for young people. For instance, poor body image is predictive of various negative outcomes, including disordered eating, low self-esteem and mood, and risky health behaviours in early adulthood, such as smoking and drug use.

Micro-interventions are designed to deliver content that aims to immediately improve specific symptoms, and they have been applied to adolescent and adult samples with body image and mood symptoms in community and digital environments. Digitally delivered micro-interventions have shown promise in improving some body image outcomes in the moment. Importantly, interactive micro-interventions that require active engagement with its content appear to be more effective than didactic or passive micro-intervention styles.

Super U intervention:

As such, this project involves the evaluation of 'Super U', a video game-based micro-intervention designed for American girls and boys. It was created in collaboration with the Dove Self-Esteem Project and Toya, a gaming studio that creates games for the Roblox platform, a hugely popular gaming platform among young people with over 57 million daily users (Roblox, September 2022). Super U is a narrative-based game, which centres around The Academy - a school for kids with superpowers - under siege by a group of rogue students bent on spreading negativity. The mission is to help players find their unique superpower of flight, fire, water, or speed, to dodge and destroy poisonous negativity to help save The Academy from being overcome. Through the engaging story of Super U, players receive messages that address known risk factors for poor body image and provide them with strategies that promote positive body image, such as learning to focus on what their body can do, instead of what it looks like; recognising that making comparisons can lead to body dissatisfaction; understanding the importance of critically evaluating messages on social media; and learning how to deal with appearance-related bullying.

Research questions:

1. Is the intervention acceptable (liked/recommended/children want to continue playing) among girls and boys in the US?
2. Is the intervention effective in eliciting immediate state-based changes in body image and mood among girls and boys in the US?
3. Is the intervention effective in eliciting short-term (one week) trait improvements in body image and related factors among girls and boys in the US?

Design:

To execute this study, the Centre for Appearance Research are collaborating with a research agency (C&R) based in the US. To test the effectiveness of Super U, we will conduct an online three-arm randomised controlled trial (RCT) among an equal number of girls and boys from a range of cities in the US.

Participants:

Recruitment will be outsourced to C&R, a US-based research agency. The research agency will recruit 90 participants for the pilot and 1479 participants for the main trial. The pilot and main trial samples will be composed of 50% girls and 50% boys, be evenly split among the age group (i.e., 9-13 years), and be representative of socioeconomic status and ethnicity. The research agency will recruit participants via their own recruitment panels of participants (children and teens) as well as through trusted and fully vetted national sample suppliers that they have successfully used in the past for research with this target group. Parental consent will be obtained.

Sample size calculations:

For the pilot, a minimum of N = 30 participants per arm (total sample N = 90) will be recruited. This recruitment objective was informed by the recommendations by Whitehead and colleagues, stating that for a main trial designed with 90% power and two-sided 5% significance, the pilot sample sizes per arm should include a minimum of 25 participants for standardised effect sizes that are expected to be small (0.2), as the ones of similar online micro-interventions have been.

For the main trial, the investigators will aim to recruit 1,479 participants (N = 493 per arm). Considering one primary outcome (state body satisfaction), and one primary end point (i.e., post-test), an a-priori power analysis based on an ANCOVA model with 3 groups and 3 covariates found that a total sample size of 967 participants would be necessary to detect small effects (F = 0.10) when considering 80% power and alpha levels of 0.05. Similar studies testing micro-interventions online show dropout rates at post-test up to 34.39%. The investigators have therefore inflated the initial sample of 967 by 35% to ensure sufficient power at post-test. Said inflation resulted in our target sample of 1479 participants, for which the investigators will aim to have a balanced distribution of gender identities and age across arms.

Procedure:

All participants will be asked to complete an online questionnaire of trait-based measures one week prior to receiving the intervention. Participants will complete these trait-based measures from their home and they will take approximately 30 minutes to complete. The questionnaires will be hosted on C&R's secure survey platform. Participants who complete the first questionnaire will then be randomised, into one of 3 groups:

1. Intervention condition: One third of participants will be randomised to receive the intervention (Super U story) described above.
2. Active control condition: One third of participants will receive an active control activity in the form of an alternative Roblox game; Rainbow Friends story which has been matched to Super U in terms of length, age appropriateness, story type and challenges.
3. Attention control condition: One third of participants will receive an attention control activity (complete word searches).

All participants will have a maximum of 30 minutes to play the game/complete word search.

Outcome measures (described in detail elsewhere):

To assess the immediate impact of playing Super U on body image and mood, all participants will complete state-based measures for body satisfaction, body functionality, and mood immediately prior to game play. At the end of game play, participants will complete the same state-based measures of body satisfaction, body functionality, and mood. Participants will also complete trait-based measures at follow up (one week after the completion of the intervention).

Other measures:

Demographics: The baseline questionnaire will capture information on age, gender, ethnicity, socio-economic status and Roblox game play frequency.

Acceptability: At post-intervention, intervention group participants will answer quantitative and qualitative questions regarding acceptability of the intervention directly following the state-based items.

Levels of engagement: At post-intervention, intervention group participants will respond to questions regarding which parts of the Super U story intervention they engaged with to track individual engagement with the active ingredients of the intervention.

Data quality measures: Items will be embedded within the surveys to assess data quality (e.g., questions to evaluate participants' attention).

Pilot study:

Initially, a pilot study will be run in the same format as the main trial (described above) with the intent to test and confirm the following to refine and validate the research design:

* Confirm recruitment strategy
* Assess the attrition rate for each phase
* Analyse acceptability data
* Assess any other elements that can help support the smooth running of the main trial
* Identify how many people engage with key elements of the game

ELIGIBILITY:
Inclusion Criteria:

* based in the United States
* aged between 9 and 13 years old
* use the Roblox gaming platform a minimum of 4 hours per week
* can read and write on their own

Exclusion Criteria:

* has played Super U Story
* do not have the written consent from a parent / caregiver to participate

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Participants who self-identify as girls or boys.
Enrollment: 2941 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-03-19 (Actual)

PRIMARY OUTCOMES:
Change in state body satisfaction (assessed via Visual Analogue Scales) | Immediately pre-intervention and immediately post-intervention
  Visual analogue scales will assess participants state level of body satisfaction. Items include: (1) "How happy do you feel about your body weight, right now?" (2) "How happy do you feel about your body shape, right now?" (3) "How happy do you feel about the way you look, right now?" Participants indicate their levels of satisfaction on a 10-point VAS (0 = extreme dissatisfaction; 10 = extreme satisfaction). A mean score across the three items will be calculated with higher scores indicating higher state body satisfaction.

SECONDARY OUTCOMES:
Change in state mood (assessed via a Visual Analogue Scale) | Immediately pre-intervention and immediately post-intervention
  A visual analogue scale will assess participants state mood using a single item. Participants will indicate their mood on a 10-point VAS (0 =very sad; 10=very happy) with higher scores indicating a more positive mood.
Change in state body functionality (assessed via a Visual Analogue Scale) | Immediately pre-intervention and immediately post-intervention
  A visual analogue scale will assess participants state body functionality using a single item 'How happy do you feel with what your body can do right now'. Participants will indicate their levels on a 10-point VAS (0 =not at all happy; 10=very happy) with higher scores indicating higher levels of body functionality.
Change in body esteem (assessed via the Body Esteem Scale for Children) | Baseline (one week prior to the intervention) and follow up (one week after the intervention is complete)
  The 20 item Body Esteem Scale for children (BES-C) assesses body esteem which refers to self-evaluations of one's body or appearance using a scale of 1 (never) to 5 (always). Once the appropriate items are reverse coded, scores on all items are averaged; with lower scores indicating lower body esteem.
Change in body appreciation (assessed via the Body Appreciation Scale -2 for Children) | Baseline (one week prior to the intervention) and follow up (one week after the intervention is complete)
  The 10 item Body Appreciation Scale-2 for Children (BAS-2C) assesses body appreciation. BAS-2C scores range from 1 (never) to 5 (always). Scores on all items are averaged; with lower scores indicating lower body appreciation.
Change in Internalisation of societal appearance ideals (assessed via the Sociocultural Attitudes Towards Appearance Questionnaire-3:General Subscale) | Baseline (one week prior to the intervention) and follow up (one week after the intervention is complete)
  The Sociocultural Attitudes Towards Appearance Questionnaire-3 (SATAQ-3): General Subscale measures internalisation of societal appearance ideals. There are 9 items from the original scale, the investigators added 3 additional items focusing specifically on social media. Scores range from 1 (totally disagree) to 5 (totally agree). Scores are averaged with higher scores indicating higher internalisation.
Change in Social media literacy (assessed via a purpose built measure) | Baseline (one week prior to the intervention) and follow up (one week after the intervention is complete)
  A 5 item purpose built measure to assess participants social media literacy, scores range from 1 (totally disagree) to 5 (totally agree) with higher scores indicating higher social media literacy.

OTHER OUTCOMES:
Total acceptability of the intervention (assessed via a self report questionnaire) | Immediately post-intervention
  Participants in the Super U intervention will complete acceptability measures via self-report questionnaire, which will include close-ended questions rated on a scale of 1 (strongly disagree) to 5 (strongly agree; e.g., I enjoyed playing Super U story) and open ended questions (e.g., What did you like about Super U Story?)
Total engagement in the intervention (assessed via a self-report questionnaire) | Immediately post-intervention
  Participants in the Super U intervention will be asked to respond to a series of questions that capture the key messages and activities they interacted with to provide a measure of intervention engagement. The response is either 'yes' or 'no' for example, 'Before traveling to the Academy, did you interact with the Selfie Guy?'

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Paraskeva, DHealth, Principal Investigator — University of the West of England
Locations (1):
- Centre for Appearance Research, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paraskeva N, Haywood S, Anquandah J, White P, Budhraja M, Diedrichs PC, Williamson H. Evaluating the Effectiveness of a Roblox Video Game (Super U Story) in Improving Body Image Among Children and Adolescents in the United States: Randomized Controlled Trial. J Med Internet Res. 2025 Jul 31;27:e66625. doi: 10.2196/66625. PMID 40743518